CLINICAL TRIAL: NCT06755073
Title: Fetal Pulmonary Artery Doppler in Mothers with Preeclampsia for Detecting Neonatal Respiratory Distress
Brief Title: Pulmonary Artery Doppler in Preeclamptic Mothers
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal M.fekry, Lecturer obstetric and gynecology, Specialist Urogynecology, Assiut University
Other Study IDs: PAD
Record Dates: First submitted 2024-12-12; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Artery Doppler
Keywords: Pulmonary Doppler; Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pulmonary artery Doppler: The four chamber view, outflow tract views, triple vessel view, longitudinal view of the aortic arch and ductal arch, and colour flow mapping will be used for a comprehensive examination to assess structural heart integrity and rule out cardiac defects. Pulmonary artery is detected and power Doppler cursor is put on it just beyond pulmonary valve and indices are calculated.
  Interventions: Radiation: Pulmonary artery Doppler ultrasound

INTERVENTIONS:
Radiation: Pulmonary artery Doppler ultrasound — Doppler ultrasound of fetal pulmonary artery

SUMMARY:
Evaluation of Pulmonary artery Doppler parameters in fetuses of mothers with severe preeclampsia

DETAILED DESCRIPTION:
Preclampsia (PE) represent a major concern in public health, affecting 2-8% of all pregnancies and considered one of the leading causes of perinatal morbidity and mortality. fetal growth restriction (FGR) ia also a common health problem affecting about 5-10% of all pregnancies and commonly associates with preeclampsia . It is estimated that 20% of cases of PE present with FGR and about 50% of early-onset FGR cases will eventually coexist with PE.

Preeclampsia affects about 5% of pregnancies and hypertensive disorders of pregnancy cause over 60,000 maternal fatalities each year around the world .The decision to deliver a woman with severe pre-eclampsia that is far from the term [mid-trimester] is difficult for the obstetrician.In most cases of highly premature pre-eclamptic gestation, certain institutions propose continuing pregnancy until one of the following occurs development of fetal lung maturity, development of fetal or maternal discomfort, or accomplishment of gestational age of 34 to 36-week of gestation .

Numerous tests have been developed in an attempt to identify if fetal lung maturation has reached a level sufficient to prevent the development of fetal RDS. These tests are based on four core themes: biochemical testing for active surfactant components, biophysical testing for surfactant functionality, physical testing of amniotic fluid opacity, and ultrasound examination of the fetuses and their tissues . Neonatal RDS has been predicted using fetal pulmonary artery Doppler. Kim and colleagues discovered that a high PAT/ET was linked to newborn RDS .The development of RDS in preterm newborns is linked to an increased acceleration time to ejection time [AT/ET] ratio in the fetal pulmonary artery .

ELIGIBILITY:
Inclusion Criteria:

* preeclampsia patients Pregnant 28 -37 weeks

Exclusion Criteria:

* fetal death Congenital fetal anomalies Fetal Cardiac arrhythmia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant woman with preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Doppler resistance index | 1 month
  Pulmonary Doppler index in fetus of preeclamptic mother

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Health Hospital, Asyut, Egypt